CLINICAL TRIAL: NCT02100345
Title: Conservative Treatment of Rectosigmoid Endometriosis Monitored by Transvaginal Ultrasound
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Bowel Endometriosis; 1-10-72-196-13 (Other: Local Ethics Committee)
Record Dates: First submitted 2014-03-21; First posted 2014-03-31 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2016-05

CONDITIONS: Bowel Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Endometriosis is a disease affecting 8-15 % of fertile women and is a cause of abdominal pain and suffering during women's menstrual periods. A subgroup of patients with DIE has an infiltration into the rectosigmoid bowel wall (4-37%). Knowledge of the growth pattern of rectosigmoid lesions related to subjective symptoms is mandatory in order to assess the need for follow-up with transvaginal ultrasound during medical treatment.

Hypotheses:

Symptoms will follow growth of rectosigmoid endometriosis.

Material and methods:

Two different cohorts of women, based on time of diagnosis of rectosigmoid endometriosis and treatment with hormonal intrauterine device or continuous oral contraceptives will receive a questionnaire and a transvaginal ultrasound scan (measuring size and volume) at inclusion, (6) and 12 months later.

Perspectives:

Patients treated conservatively may be followed by questionnaires, thereby reducing the need for time consuming clinical controls.

ELIGIBILITY:
Inclusion Criteria:

* Medically treated bowel endometriosis

Exclusion Criteria:

* Age below 18 years
* Bowel resection of any kind
* Cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with bowel endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Transvaginal Ultrasound | 29 months

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Mr Seyer-Hansen, MD, PhD, Study Director — Department of Obstetrics and Gynecology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Region Midt, Denmark